CLINICAL TRIAL: NCT03966040
Title: A Single-center, Open-label, Phase Ib Clinical Trial to Evaluate the Safety and Immunogenicity of a Recombinant Staphylococcus Aureus Vaccine (Escherichia Coli) With Different Dose in Healthy Adults Aged 18-70 Years in China
Brief Title: A Clinical Trial to Evaluate a Recombinant Staphylococcus Aureus Vaccine (Escherichia Coli) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Chengdu Olymvax Biopharmaceuticals Inc. (Industry); PLA Army Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT049
Record Dates: First submitted 2019-05-25; First posted 2019-05-29 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2019-05

CONDITIONS: Staphylococcus Aureus Infection
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immunization schedule of day 0-3-7 (Experimental): Three doses of schedule given at day 0, 3 and 7.
  Interventions: Biological: Inoculate Staphylococcus aureus vaccine(Escherichia Coli) at day 0-3-7
- Immunization schedule of day 0/0-3-7 (Experimental): Four doses of schedule given at day 0/0, 3 and 7.
  Interventions: Biological: Inoculate Staphylococcus aureus vaccine(Escherichia Coli) at day 0/0-3-7
- Immunization schedule of day 0/0-7 (Experimental): Three doses of schedule given at day 0/0 and 7.
  Interventions: Biological: Inoculate Staphylococcus aureus vaccine(Escherichia Coli) at day 0/0-7
- Immunization schedule of day 0/0-7-14 (Experimental): Four doses of schedule given at day 0/0, 7 and 14.
  Interventions: Biological: Inoculate Staphylococcus aureus vaccine(Escherichia Coli) at day 0/0-7-14

INTERVENTIONS:
Biological: Inoculate Staphylococcus aureus vaccine(Escherichia Coli) at day 0-3-7 — 36 participants will be given three dose of Staphylococcus aureus vaccine(Escherichia Coli) at day 0-3-7
  Arms: Immunization schedule of day 0-3-7
Biological: Inoculate Staphylococcus aureus vaccine(Escherichia Coli) at day 0/0-3-7 — 36 participants will be given four dose of Staphylococcus aureus vaccine(Escherichia Coli) at day 0/0-3-7
  Arms: Immunization schedule of day 0/0-3-7
Biological: Inoculate Staphylococcus aureus vaccine(Escherichia Coli) at day 0/0-7 — 36 participants will be given three dose of Staphylococcus aureus vaccine(Escherichia Coli) at day 0/0-7
  Arms: Immunization schedule of day 0/0-7
Biological: Inoculate Staphylococcus aureus vaccine(Escherichia Coli) at day 0/0-7-14 — 36 participants will be given four dose of Staphylococcus aureus vaccine(Escherichia Coli) at day 0/0-7-14
  Arms: Immunization schedule of day 0/0-7-14

SUMMARY:
This is a single center, open-label phase1b clinical trial. The study will evaluate the safety and immunogenicity of an experimental recombinant staphylococcus aureus vaccine with different immunization schedules in healthy adults aged 18-70 years, including day 0-3-7, day 0/0-3-7, day 0/0-7 and day 0/0-7-14.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 70 years (aged over 18 and under 71 years)

  * Able to comply with all clinical trial protocol requirements and willing to complete all the visit plan process during the whole clinical trial observation period.
  * Able to understand the content of informed consent and willing to sign the informed consent.
  * Able to complete the diary card independently.
  * For females only (18-49 years), a negative urine pregnancy test and willing to practice continuous effective contraception during the study.
  * Axillary temperature ≤37.0°C.

Exclusion Criteria:

* • Prior receipt of Staphylococcus aureus vaccine

  * Any confirmed Staphylococcus aureus infection disease in the past 12 month.
  * History of asthma, hereditary angioneurotic edema, diabetes, malignancy or other serious disease. Participation in the clinical trial is likely to increase the disease risk and interfere with the observation of clinical trial index.
  * Prior blood donation or Blood loss over 400ml in the last 3 months;
  * Coagulation disorders (coagulation factor deficiency, coagulopathy or platelet disorder) diagnosed by doctors, or obvious bruises or blood coagulation noticed.
  * History of allergic disease likely to be exacerbated by any component of the vaccine, including allergy, urticaria, respiratory difficulty, angioneurotic edema or abdominal pain. Any autoimmune disease or immunodeficient state, parents, brother and sister with autoimmune disease or immunodeficient disease.
  * Taking immunoglobulins and/or any blood products within the last 12 months.
  * Asplenia, functional asplenia or asplenia caused by any situation or splenectomy.
  * Any acute disease or acute attack of chronic disease in last 7 days.
  * History of thyroidectomy or thyroid disease requiring treatment in the last 12 months.
  * Immunosuppressor, cytotoxic therapy, inhaled corticosteroid (excluding corticosteroids spray treatment of allergic rhinitis, acute and nonconcurrent corticosteroids treatment)
  * Participation in another research study involving receipt of an investigational product in the last 30 days.
  * Woman who is breast-feeding.
  * Prior administration of attenuated vaccine in last 28 days.
  * Prior administration of subunit vaccine, inactivated vaccine or allergic therapy in last 14 days.
  * Current anti-tuberculosis therapy or HIV infected individuals
  * Any other conditions may compromise the safety or availability of participants in the judgment of the investigator.

Following Immunization exclusion standard:

* Other condition violates the inclusion criteria or meets the exclusion criteria is noticed after the first immunization.
* Any grade 3 or more serious adverse reaction associated with vaccination since the last vaccination.
* According to the investigator, the participant should not continue participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited adverse reactions after vaccination | within 21 days after vaccination
  Occurrence of solicited adverse reactions within 21 days afte vaccination with the Recombinant

SECONDARY OUTCOMES:
Occurrence of unsolicited adverse reactions after vaccination | within 42 days after the vaccination
  Occurrence of unsolicited adverse reactions within 42 days after vaccination with the Recombinant Staphylococcus aureus vaccine
Occurrence of serious adverse events after the vaccination. | within 6 months after the vaccination
  Occurrence of serious adverse events within 6 months after the vaccination with the Recombinant Staphylococcus aureus vaccine
Changes of the blood routine after vaccination. | within 17 days after the vaccination
  Changes of the blood routine after vaccination with the Recombinant Staphylococcus aureus vaccine on day 3, 7, 10, 14 and 17.
Changes of the blood biochemistry after vaccination. | within 17 days after the vaccination
  Changes of the blood biochemistry after vaccination with the Recombinant Staphylococcus aureus vaccine on day 3, 7, 10, 14 and 17.
Antibody responses against 5 specific antigens in Staphylococcus aureus vaccine | within 42 days after vaccianation
  Antibody responses against 5 specific antigens in Staphylococcus aureus vaccine at day 7, 14, 21 and 42, respectively.
Specific functional antibody responses to the Staphylococcus aureus vaccine | within 42 days after vaccianation
  Specific functional antibody responses to the Staphylococcus aureus vaccine at day 7, 14, 21 and 42

CONTACTS AND LOCATIONS:
Overall Officials: Fangyue Meng, Master, Study Director — Jiangsu, China
Locations (1):
- Suining County Center for Disease Control and Prevention, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data for all primary and secondary outcomes will be made available within 6 months of study completion.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: within 6 months of study completion
Access Criteria: Data access requests will be reviewed by the sponsor and requestors will be required to sign a Date Access Agreement.

REFERENCES:
- [Derived] Zhu FC, Zeng H, Li JX, Wang B, Meng FY, Yang F, Gu J, Liang HY, Hu YM, Liu P, Peng LS, Hu XK, Zhuang Y, Fan M, Li HB, Tan ZM, Luo P, Zhang P, Chu K, Zhang JY, Zeng M, Zou QM. Evaluation of a recombinant five-antigen Staphylococcus aureus vaccine: The randomized, single-centre phase 1a/1b clinical trials. Vaccine. 2022 May 20;40(23):3216-3227. doi: 10.1016/j.vaccine.2022.04.034. Epub 2022 Apr 23. PMID 35473663
- [Derived] Wei J, Cheng X, Zhang Y, Gao C, Wang Y, Peng Q, Luo P, Yang L, Zou Q, Zeng H, Gu J. Identification and application of a neutralizing epitope within alpha-hemolysin using human serum antibodies elicited by vaccination. Mol Immunol. 2021 Jul;135:45-52. doi: 10.1016/j.molimm.2021.03.028. Epub 2021 Apr 16. PMID 33873093